CLINICAL TRIAL: NCT04026256
Title: Mechanisms Underlying the Bone Modeling Effects of Combined Anabolic/Antiresorptive Administration
Brief Title: Bone Modeling Effects of Combined Anabolic/Antiresorptive Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018P002537; 5R01AR073191-04 (NIH)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Postmenopausal Osteoporosis
Keywords: osteoporosis; histomorphometry; bone density; teriparatide; denosumab
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Teriparatide; Denosumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Teriparatide only (Active Comparator): daily subcutaneous injection teriparatide for 3 months
  Interventions: Drug: Teriparatide
- Denosumab only (Active Comparator): one dose of subcutaneous injection denosumab
  Interventions: Drug: Denosumab
- Denosumab and teriparatide (Active Comparator): daily subcutaneous injection teriparatide for 3 months plus one dose of subcutaneous injection denosumab
  Interventions: Drug: Teriparatide; Drug: Denosumab

INTERVENTIONS:
Drug: Teriparatide — teriparatide daily subcutaneous injection
  Other Names: Forteo
  Arms: Denosumab and teriparatide; Teriparatide only
Drug: Denosumab — denosumab subcutaneous injection
  Other Names: Prolia
  Arms: Denosumab and teriparatide; Denosumab only

SUMMARY:
The purpose of this study is to examine, via iliac crest bone biopsies, the mechanism of combined teriparatide and denosumab on the bone of postmenopausal osteoporotic women after 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* women aged 45+
* postmenopausal
* osteoporotic with high risk of fracture

Exclusion Criteria:

* significant previous use of bone health modifying treatments
* known congenital or acquired bone disease other than osteoporosis
* significant renal disease, liver disease, cardiopulmonary disease, or psychiatric disease
* abnormal calcium or parathyroid hormone level
* serum vitamin D <20 ng/mL or >60ng/mL
* serum alkaline phosphatase above upper normal limit with no explanation
* anemia (hematocrit <32%)
* history of malignancy (except non-melanoma skin carcinoma), radiation therapy, or gouty arthritis
* history of urolithiasis within the last one year
* excessive alcohol use or substance abuse
* use of oral or parenteral glucocorticoids for more than 14 days within the past 6 months
* extensive dental work involving extraction or dental implant within the past or upcoming 2 months
* known sensitivity to mammalian cell-derived drug products
* known contraindications to denosumab, teriparatide, or any of their excipients
* known contraindications to tetracycline, demeclocycline, or other antibiotics in this drug class
* continuous use of tetracycline for >1-month duration within the last 10 years

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Leder, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 participants enrolled in the study. 3 participants withdrew their consent very soon after signing the consent form and PRIOR to randomization to a treatment arm. Thus we are reporting this as 37 enrolled in the study and 34 enrolled AND randomized.
Period: Overall Study
Arm/Group | Teriparatide Only | Denosumab Only | Denosumab and Teriparatide
Started | 13 | 9 | 12
Completed | 10 | 8 | 9
Not Completed | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: refers to subjects enrolled and randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide Only | Denosumab Only | Denosumab and Teriparatide | Total
Number analyzed (Participants) | 13 | 9 | 12 | 34
Age, Continuous [Mean (Full Range); unit: years] | 66 [50 to 79] | 64 [55 to 71] | 65 [55 to 72] | 66 [50 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 12 | 34
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 12 | 8 | 11 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 3 | 5
  White | 10 | 8 | 8 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Lumbar Spine bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DXA) (g/cm2) [Mean (Standard Deviation); unit: g/cm2] | 0.87 (0.09) | 0.80 (0.09) | 0.81 (0.06) | 0.83 (0.08)
Femoral Neck BMD by DXA (g/cm2) [Mean (Standard Deviation); unit: g/cm2] | 0.62 (0.07) | 0.64 (0.06) | 0.60 (0.08) | 0.62 (0.07)
Total Hip BMD by DXA (g/cm2) [Mean (Standard Deviation); unit: g/cm2] | 0.75 (0.11) | 0.73 (0.08) | 0.72 (0.10) | 0.74 (0.10)

OUTCOME MEASURES:

1. Primary Outcome: Cancellous Bone Formation Rate at Month 3
Description: Cancellous bone formation rate at month 3 is calculated from the cancellous (trabecular) compartment of the iliac crest bone biopsy specimens.
  Bone formation rate (BFR/BS, mm3/mm2/day): amount of new bone formed in unit time per unit of bone surface. It is calculated by multiplying the mineralizing surface/bone surface (MS/BS) by the mineral apposition rate (MAR) - see below for how MS/BS and MAR are calculated.
  Mineralizing surface (MS/BS, %): is the percent of bone surface that displays a tetracycline label reflecting active mineralization. It is calculated as the double-labeled surface plus one half of the single-labeled surface and is expressed as a function of total bone surface. It is a measure of the proportion of bone surface upon which new mineralized bone was being deposited during the period of tetracycline labeling.
  Mineral apposition rate (MAR mm/day): is the mean distance between the double labels, divided by the time interval between them.
Time Frame: 3 months after first dose of study drug
Population: refers to number of subjects who had bone biopsies available for analysis.
Measure: Mean (Standard Deviation); unit: mm3/mm2/day
Arm/Group | Teriparatide Only | Denosumab Only | Denosumab and Teriparatide
Number analyzed (Participants) | 9 | 8 | 9
mm3/mm2/day | 0.13 (0.06) | 0.01 (0.01) | 0.06 (0.02)

ADVERSE EVENTS:
Time Frame: adverse event data was collected from baseline to approximately 1 month after study completion, for an average duration of 5 months per participant (assuming that the participant completed the whole study).
Arm/Group | Teriparatide Only | Denosumab Only | Denosumab and Teriparatide
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/9 | 1/12
Other Adverse Events (participants affected / at risk) | 5/13 | 6/9 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teriparatide Only (N=13) | Denosumab Only (N=9) | Denosumab and Teriparatide (N=12)
phototoxic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — phototoxic dermatitis likely secondary to demeclocycline used for biopsy labelling
transient syncopal event (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Teriparatide Only (N=13) | Denosumab Only (N=9) | Denosumab and Teriparatide (N=12)
rhinorrhea (Ear and labyrinth disorders) | 2 | 1 | 2
nausea (Gastrointestinal disorders) | 4 | 2 | 4
joint pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
propagation of fracture at biopsy site (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
dizziness (Nervous system disorders) | 1 | 1 | 2
headache (Nervous system disorders) | 2 | 0 | 4
pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
fatigue (General disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT04026256/Prot_SAP_000.pdf